CLINICAL TRIAL: NCT01014585
Title: A Multicenter, Randomized, Double-blind, Placebo-Controlled Discontinuation Study of the Durability of Effect of Milnacipran for the Treatment of Fibromyalgia in Patients Receiving Long-term Milnacipran Treatment
Brief Title: Discontinuation Study of the Durability of Effect of Milnacipran for the Treatment of Fibromyalgia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Forest Laboratories (Industry)
Collaborators: Cypress Bioscience, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MLN-MD-27
Record Dates: First submitted 2009-11-13; First posted 2009-11-17 (Estimated); Results first posted 2011-09-07 (Estimated); Last update posted 2011-09-07 (Estimated); Status verified 2011-09

CONDITIONS: Fibromyalgia
Keywords: Milnacipran; Pain; Durability of Effect; Loss of Therapeutic Response; Fatigue; Forest Research Institute; Savella ®
MeSH Terms: conditions — Fibromyalgia; Pain; Fatigue | interventions — Milnacipran

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Placebo Comparator): Placebo tablets administered orally twice daily
  Interventions: Drug: Placebo
- 2 (Experimental): Milnacipran tablets administered orally twice daily
  Interventions: Drug: Milnacipran

INTERVENTIONS:
Drug: Placebo — Placebo tablets administered orally twice daily
  Arms: 1
Drug: Milnacipran — Milnacipran tablets administered orally twice daily
  Other Names: Savella ®
  Arms: 2

SUMMARY:
The purpose of this study is to evaluate the durability of effect of milnacipran for the treatment of fibromyalgia in patients receiving long-term milnacipran treatment and to characterize the effects of milnacipran on multiple symptoms of fibromyalgia, as demonstrated by changes in symptoms following the discontinuation of milnacipran.

ELIGIBILITY:
Inclusion Criteria:

* Currently participating in Study MLN-MD-06
* Receiving a stable dosage of milnacipran (50-200 mg/d) at Screening/Enrollment (Visit 1)

Exclusion Criteria:

* Significant risk of suicide
* History of mania, bipolar disorder, psychotic disorder, schizophrenia, or a current episode of major depressive disorder
* Myocardial infarction and/or stroke within the prior 12 months
* Mean systolic blood pressure > 180 mm Hg or mean diastolic blood pressure > 110 mm Hg at Screening (Visit 1)
* Active liver disease
* Severe renal impairment
* Platelet and bleeding disorders
* Female patients who are pregnant or breastfeeding

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 340 (Actual)
Dates: Start 2009-11; Primary Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joel Trugman, MD, Study Director — Forest Research Institute Inc., A Subsidiary of Forest Laboratories Inc
Locations (58):
- United States (58):
  - Forest Investigative Site 062, Birmingham, Alabama
  - Forest Investigative Site 065, Birmingham, Alabama
  - Forest Investigative Site 012, Tucson, Arizona
  - Forest Investigative Site 007, Fresno, California
  - Forest Investigative Site 032, Pismo Beach, California
  - Forest Investigative Site 025, Sacramento, California
  - Forest Investigative Site 019, San Diego, California
  - Forest Investigative Site 057, Santa Ana, California
  - Forest Investigative Site 039, Vista, California
  - Forest Investigative Site 050, Cromwell, Connecticut
  - Forest Investigative Site 049, Danbury, Connecticut
  - Forest Investigative Site 055, Stamford, Connecticut
  - Forest Investigative Site 011, Delray Beach, Florida
  - Forest Investigative Site 013, Ocala, Florida
  - Forest Investigative Site 016, Orlando, Florida
  - Forest Investigative Site 043, Palm Harbor, Florida
  - Forest Investigative Site 060, Pembroke Pines, Florida
  - Forest Investigative Site 066, Atlanta, Georgia
  - Forest Investigative Site 009, Atlanta, Georgia
  - Forest Investigative Site 026, Honolulu, Hawaii
  - Forest Investigative Site 056, Libertyville, Illinois
  - Forest Investigative Site 038, Peoria, Illinois
  - Forest Investigative Site 031, Evansville, Indiana
  - Forest Investigative Site 064, Frederick, Maryland
  - Forest Investigative Site 030, Newton, Massachusetts
  - Forest Investigative Site 048, North Dartmouth, Massachusetts
  - Forest Investigative Site 017, Springfield, Massachusetts
  - Forest Investigative Site 008, Worcester, Massachusetts
  - Forest Investigative Site 061, Kalamazoo, Michigan
  - Forest Investigative Site 020, Jackson, Mississippi
  - Forest Investigative Site 004, St Louis, Missouri
  - Forest Investigative Site 033, Cherry Hill, New Jersey
  - Forest Investigative Site 040, Albuquerque, New Mexico
  - Forest Investigative Site 035, Great Neck, New York
  - Forest Investigative Site 014, Rochester, New York
  - Forest Investigative Site 027, Syracuse, New York
  - Forest Investigative Site 054, Charlotte, North Carolina
  - Forest Investigative Site 018, Greensboro, North Carolina
  - Forest Investigative Site 002, Greenville, North Carolina
  - Forest Investigative Site 024, Salisbury, North Carolina
  - Forest Investigative Site 042, Winston-Salem, North Carolina
  - Forest Investigative Site 003, Cincinnati, Ohio
  - Forest Investigative Site 005, Cleveland, Ohio
  - Forest Investigative Site 059, Columbus, Ohio
  - Forest Investigative Site 044, Eugene, Oregon
  - Forest Investigative Site 010, Eugene, Oregon
  - Forest Investigative Site 001, Medford, Oregon
  - Forest Investigative Site 052, Medford, Oregon
  - Forest Investigative Site 041, Portland, Oregon
  - Forest Investigative Site 051, Duncansville, Pennsylvania
  - Forest Investigative Site 046, Mechanicsburg, Pennsylvania
  - Forest Investigative Site 028, Anderson, South Carolina
  - Forest Investigative Site 021, Greer, South Carolina
  - Forest Investigative Site 006, Salt Lake City, Utah
  - Forest Investigative Site 015, Chesapeake, Virginia
  - Forest Investigative Site 047, Seattle, Washington
  - Forest Investigative Site 036, Wenatchee, Washington
  - Forest Investigative Site 063, Racine, Wisconsin

REFERENCES:
- [Derived] Clauw DJ, Mease PJ, Palmer RH, Trugman JM, Wang Y. Continuing efficacy of milnacipran following long-term treatment in fibromyalgia: a randomized trial. Arthritis Res Ther. 2013 Aug 16;15(4):R88. doi: 10.1186/ar4268. PMID 23953493

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period was from November 2009 through February 2010 at 58 centers in the United States with the last patient visit occurring on June 7, 2010.
Pre-assignment Details: Upon completion of a long term milnacipran open label study MLN-MD-06, patients were enrolled in the current study MLN-MD-27 (NCT01014585), and received open label treatment with milnacipran for four weeks prior to randomization.
Groups:
- Responders: Placebo (Milnacipran Withdrawn); Responders: Milnacipran (Milnacipran Continued): The Randomized Population for Responders
- Non-Responders: Placebo (Milnacipran Withdrawn); Non-Responders: Milnacipran (Milnacipran Continued): The Randomized Population for Non-Responders
Period: Overall Study
Arm/Group | Responders: Placebo (Milnacipran Withdrawn) | Responders: Milnacipran (Milnacipran Continued) | Non-Responders: Placebo (Milnacipran Withdrawn) | Non-Responders: Milnacipran (Milnacipran Continued)
Started | 51 | 100 | 60 | 129
Completed | 31 | 75 | 37 | 99
Not Completed | 20 | 25 | 23 | 30
Not completed — Adverse Event | 0 | 2 | 0 | 3
Not completed — Withdrawal by Subject | 2 | 0 | 1 | 3
Not completed — Lost to Follow-up | 0 | 0 | 0 | 2
Not completed — Withdrawn Due to Worsening Fibromyalgia | 18 | 23 | 22 | 22

BASELINE CHARACTERISTICS:
Groups:
- Responders: Placebo (Milnacipran Withdrawn): Safety Population for Responders: placebo treatment assignment
  One patient in the randomized population for responders assigned to placebo did not take at least one dose of double blind investigational product and therefore was not included in the Safety Population.
- Responders: Milnacipran (Milnacipran Continued): Safety Population for Responders: milnacipran treatment assignment
- Non-Responders: Placebo (Milnacipran Withdrawn): Safety Population for Non-Responders: placebo treatment assignment
- Non-Responders: Milnacipran (Milnacipran Continued): Safety Population for Non-Responders: milnacipran treatment assignment
  One patient in the randomized population for non-responders assigned to milnacipran did not take at least one dose of double-blind investigational product and therefore was not included in the Safety population.
- Total: Total of all reporting groups
Arm/Group | Responders: Placebo (Milnacipran Withdrawn) | Responders: Milnacipran (Milnacipran Continued) | Non-Responders: Placebo (Milnacipran Withdrawn) | Non-Responders: Milnacipran (Milnacipran Continued) | Total
Number analyzed (Participants) | 50 | 100 | 60 | 128 | 338
Age Continuous [Mean (Standard Deviation); unit: years] | 54.0 (8.3) | 54.5 (9.3) | 54.7 (9.6) | 54.8 (9.4) | 54.6 (9.2)
Age, Customized [Number; unit: Years]
  Between 20 and 60 years | 39 | 73 | 38 | 86 | 236
  >=60 years | 11 | 27 | 22 | 42 | 102
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 96 | 59 | 122 | 325
  Male | 2 | 4 | 1 | 6 | 13
Region of Enrollment [Number; unit: participants]
  United States | 50 | 100 | 60 | 128 | 338

OUTCOME MEASURES:

1. Primary Outcome: Time to Loss of Therapeutic Response (LTR)
Description: Time to loss of therapeutic response is defined as the time from the first dose of double-blind investigational product to the first visit when a patient has a < 30% reduction in Visual Analog Scale (VAS) pain score from pre-milnacipran exposure OR a worsening of fibromyalgia requiring, in the judgment of the investigator, an alternative treatment
Time Frame: From baseline Visit 3 (week 5) to Visit 7 (week 17)
Population: The Intent to Treat (ITT) Population for Responders is defined as all patients in the Safety Population for Responders with at least 1 post-baseline assessment of primary efficacy parameter. All patients in the Safety Population were included in the ITT population. No efficacy statistical analyses were performed for the Non-Responder population.
Measure: Median (95% Confidence Interval); unit: Days
Groups:
- Responders: Placebo (Milnacipran Withdrawn): Intent to Treat (ITT) Population for Responders: placebo treatment assignment, matching placebo administered orally twice per day.
- Responders: Milnacipran (Milnacipran Continued): Intent to Treat (ITT) Population for Responders: milnacipran treatment assignment, milnacipran 50-200 mg per day, administered orally twice per day.
- Non-Responders: Placebo (Milnacipran Withdrawn): Intent to Treat (ITT) Population for Non-Responders: placebo treatment assignment, matching placebo, administered orally twice per day.
- Non-Responders: Milnacipran (Milnacipran Continued): Intent to Treat (ITT) Population for Non-Responders: milnacipran treatment assignment, 50-200 mg per day, administered orally twice per day.
Arm/Group | Responders: Placebo (Milnacipran Withdrawn) | Responders: Milnacipran (Milnacipran Continued) | Non-Responders: Placebo (Milnacipran Withdrawn) | Non-Responders: Milnacipran (Milnacipran Continued)
Number analyzed (Participants) | 50 | 100 | 0 | 0
Days | 56 [28 to 85] | NA [NA to NA] — NA represents not estimable. Not enough participants experienced a loss of therapeutic response to calculate the median value and 95 percent confidence interval. |  |
Statistical Analysis 1: Comparison: Responders: Placebo (Milnacipran Withdrawn) vs Responders: Milnacipran (Milnacipran Continued); Test type: Superiority or Other; p = 0.0004, Log Rank; Hazard Ratio (HR) = 0.44, 95% CI 2-sided [0.27 to 0.71]
Statistical Analysis 2: Comparison: Responders: Placebo (Milnacipran Withdrawn); Test type: Superiority or Other; Days until LTR at the 25th percentile = 18
Statistical Analysis 3: Comparison: Responders: Milnacipran (Milnacipran Continued); Test type: Superiority or Other; Days until LTR at the 25th percentile = 45

2. Secondary Outcome: Time to Worsening in Patient Global Impression of Change (PGIC)
Description: Time to worsening in Patient Global Impression of Change is defined as the time from the first dose of double-blind investigational product to the first visit when a patient has a PGIC score of 6 or 7. The PGIC is an efficacy assessment on a scale of 1-7 taken at visits 4, 5, 6 and 7. The wording of the assessment is as follows: "Since the start of the study, overall my fibromyalgia is:" 1=Very Much Improved, 2=Much Improved, 3=Minimally Improved, 4=No Change, 5=Minimally Worse, 6=Much Worse, and 7=Very Much Worse.
Time Frame: From baseline Visit 3 (week 5) to Visit 7 (week 17)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Responders: Placebo (Milnacipran Withdrawn) | Responders: Milnacipran (Milnacipran Continued) | Non-Responders: Placebo (Milnacipran Withdrawn) | Non-Responders: Milnacipran (Milnacipran Continued)
Number analyzed (Participants) | 50 | 100 | 0 | 0
Days | 86 [30 to NA] — NA represents not estimable. Not enough participants experienced a worsening in PGIC to calculate the upper bound of 95 percent confidence interval. | NA [NA to NA] — NA represents not estimable. Not enough participants experienced a worsening in PGIC to calculate the median value and the 95 percent confidence interval. |  |
Statistical Analysis 1: Comparison: Responders: Placebo (Milnacipran Withdrawn) vs Responders: Milnacipran (Milnacipran Continued); Test type: Superiority or Other; p = 0.0002, Log Rank; Hazard Ratio (HR) = 0.36, 95% CI 2-sided [0.20 to 0.63]
Statistical Analysis 2: Comparison: Responders: Placebo (Milnacipran Withdrawn); Test type: Superiority or Other; Days until LTR at the 25th percentile = 22

3. Secondary Outcome: Time to Worsening in Multidimensional Assessment of Fatigue (MAF)
Description: Time to worsening in MAF is defined as the time from the first dose of double-blind investigational product to the first visit when a patient has a 10-point increase from baseline in the global index of fatigue in MAF. Scores range from 1 (no fatigue) to 50 (severe fatigue). The MAF contains 16 items measuring 4 dimensions of fatigue: severity, distress, degree of interference in activities of daily living, and timing. Fourteen of the items contain numerical rating scales (increasing in severity); the remaining 2 items have multiple-choice responses (decreasing in severity).
Time Frame: From baseline Visit 3 (week 5) to Visit 7 (week 17)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Responders: Placebo (Milnacipran Withdrawn) | Responders: Milnacipran (Milnacipran Continued) | Non-Responders: Placebo (Milnacipran Withdrawn) | Non-Responders: Milnacipran (Milnacipran Continued)
Number analyzed (Participants) | 50 | 100 | 0 | 0
Days | NA [NA to NA] — NA represents not estimable. Not enough participants experienced a worsening in the MAF to calculate the median value and the 95 percent confidence interval. | NA [NA to NA] — NA represents not estimable. Not enough participants experienced a worsening in the MAF to calculate the median value and the 95 percent confidence interval. |  |
Statistical Analysis 1: Comparison: Responders: Placebo (Milnacipran Withdrawn) vs Responders: Milnacipran (Milnacipran Continued); Test type: Superiority or Other; p = 0.4104, Log Rank; Hazard Ratio (HR) = 0.80, 95% CI 2-sided [0.46 to 1.38]
Statistical Analysis 2: Comparison: Responders: Placebo (Milnacipran Withdrawn); Test type: Superiority or Other; Days until LTR at the 25th percentile = 18
Statistical Analysis 3: Comparison: Responders: Milnacipran (Milnacipran Continued); Test type: Superiority or Other; Days until LTR at the 25th percentile = 30

ADVERSE EVENTS:
Groups:
- Non-Responders: Milnacipran (Milnacipran Continued): Safety Population for Non-Responders: milnacipran treatment assignment
  One patient in the randomized population for non-responders assigned to milnacipran did not take at least one dose of double blind investigational product and therefore was not included in the Safety population.
Arm/Group | Responders: Placebo (Milnacipran Withdrawn) | Responders: Milnacipran (Milnacipran Continued) | Non-Responders: Placebo (Milnacipran Withdrawn) | Non-Responders: Milnacipran (Milnacipran Continued)
Serious Adverse Events (participants affected / at risk) | 0/50 | 1/100 | 1/60 | 3/128
Other Adverse Events (participants affected / at risk) | 8/50 | 6/100 | 10/60 | 30/128
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Responders: Placebo (Milnacipran Withdrawn) (N=50) | Responders: Milnacipran (Milnacipran Continued) (N=100) | Non-Responders: Placebo (Milnacipran Withdrawn) (N=60) | Non-Responders: Milnacipran (Milnacipran Continued) (N=128)
Non-cardiac chest pain (General disorders) | 0 | 1 | 0 | 0
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 0 | 1
Hidradenitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Responders: Placebo (Milnacipran Withdrawn) (N=50) | Responders: Milnacipran (Milnacipran Continued) (N=100) | Non-Responders: Placebo (Milnacipran Withdrawn) (N=60) | Non-Responders: Milnacipran (Milnacipran Continued) (N=128)
Sinusitis (Infections and infestations) | 3 | 4 | 1 | 11
Oedema peripheral (General disorders) | 3 | 2 | 1 | 0
Irritability (General disorders) | 3 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 4 | 1 | 9
Upper respiratory tract infection (Infections and infestations) | 2 | 4 | 1 | 7
Nausea (Gastrointestinal disorders) | 1 | 4 | 3 | 4
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 1 | 3 | 3 | 3
Bronchitis (Infections and infestations) | 1 | 2 | 3 | 2
Constipation (Gastrointestinal disorders) | 0 | 2 | 3 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All data generated in this study is the property of Forest Research Institute, Inc. An integrated clinical and statistical report was prepared at the completion of the study. Publication of the results by the Investigator will be subject to mutual agreement between the Investigator and Forest Research Institute, Inc.